CLINICAL TRIAL: NCT04795479
Title: A Randomized, Partial Double-Blind, Placebo- and Positive- Controlled, Multiple-Dose, 4-Way Crossover, Thorough QT/QTc (TQT) Study to Investigate the Effect of Relacorilant on Cardiac Repolarization in Healthy Volunteers
Brief Title: T/QT Study to Investigate the Effect of Relacorilant on Cardiac Repolarization in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CORT125134-130
Record Dates: First submitted 2021-01-29; First posted 2021-03-12 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Treatment Sequence 1 (Experimental): Participants will receive relacorilant 400 mg once daily (QD) for 5 days in Period 1, followed by relacorilant 800 mg QD for 5 days in Period 2, followed by placebo to relacorilant QD for 5 days in Period 3, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 2 (Experimental): Participants will receive relacorilant 800 mg QD for 5 days in Period 1, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 2, followed by relacorilant 400 mg QD for 5 days in Period 3, followed by placebo to relacorilant QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 3 (Experimental): Participants will receive placebo to relacorilant QD for 5 days in Period 1, followed by relacorilant 400 mg QD for 5 days in Period 2, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 3, followed by relacorilant 800 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 4 (Experimental): Participants will receive relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 1, followed by placebo to relacorilant QD for 5 days in Period 2, followed by relacorilant 800 mg QD for 5 days in Period 3, followed by relacorilant 400 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 5 (Experimental): Participants will receive relacorilant 800 mg QD for 5 days in Period 1, followed by placebo to relacorilant QD for 5 days in Period 2, followed by relacorilant 400 mg QD for 5 days in Period 3, followed by relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 6 (Experimental): Participants will receive placebo to relacorilant QD for 5 days in Period 1, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 2, followed by relacorilant 800 mg QD for 5 days in Period 3, followed by relacorilant 400 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 7 (Experimental): Participants will receive relacorilant 400 mg QD for 5 days in Period 1, followed by relacorilant 800 mg QD for 5 days in Period 2, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 3, followed by placebo to relacorilant QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 8 (Experimental): Participants will receive placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 1, followed by relacorilant 400 mg QD for 5 days in Period 2, followed by placebo to relacorilant QD for 5 days in Period 3, followed by relacorilant 800 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 9 (Experimental): Participants will receive placebo to relacorilant QD for 5 days in Period 1, followed by relacorilant 400 mg QD for 5 days in Period 2, followed by relacorilant 800 mg QD for 5 days in Period 3, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 10 (Experimental): Participants will receive relacorilant 400 mg QD for 5 days in Period 1, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 2, followed by placebo to relacorilant QD for 5 days in Period 3, followed by relacorilant 800 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 11 (Experimental): Participants will receive relacorilant 800 mg QD for 5 days in Period 1, followed by placebo to relacorilant QD for 5 days in Period 2, followed by placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 3, followed by relacorilant 400 mg QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin
- Treatment Sequence 12 (Experimental): Participants will receive placebo to relacorilant QD for 4 days and moxifloxacin 400 mg on Day 5 in Period 1, followed by relacorilant 800 mg QD for 5 days in Period 2, followed by relacorilant 400 mg QD for 5 days in Period 3, followed by placebo to relacorilant QD for 5 days in Period 4. Treatment periods will be separated by a washout of at least 10 days.
  Interventions: Drug: Relacorilant; Drug: Placebo to relacorilant; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Relacorilant — Relacorilant 400 mg (therapeutic dose) or 800 mg (supra-therapeutic dose) capsule by mouth once daily
  Other Names: CORT125134
Drug: Placebo to relacorilant — Placebo to relacorilant capsule by mouth once daily
Drug: Moxifloxacin — Moxifloxacin 400 mg tablet by mouth

SUMMARY:
This dedicated T/QT study will investigate the effect of relacorilant on cardiac repolarization in healthy participants.

DETAILED DESCRIPTION:
This four-period crossover study with 12 treatment sequences includes relacorilant administered at therapeutic (400 mg once daily [QD]) and supra-therapeutic (800 mg QD) doses, placebo for relacorilant as a negative control, and oral moxifloxacin as a positive control. The positive control will serve to determine the sensitivity of the assay to detect small increases from baseline in the QTc interval. Each of the four treatment periods will last 5 days with a washout of at least 10 days between periods. Relacorilant and placebo to relacorilant will be administered double-blind; moxifloxacin will be administered open label.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a BMI ≥18.0 kg/m^2 and ≤30.0 kg/m^2 at screening
* No clinically significant abnormal findings with the physical examination, medical/surgical/medication history, vital signs, or clinical laboratory assessments and adequate cardiac conduction by electrocardiogram (ECG) without evidence of first-, second- or third-degree atrioventricular block
* Female participants of childbearing potential with a negative serum pregnancy test at screening and urine pregnancy test on Day -1 of Period 1
* All male participants agree to use condom to prevent exposure to partner; male participants with female partner of childbearing potential to use a second method of contraception
* Female participants of childbearing potential agree to use the highly effective contraception of low user dependency
* Participant is willing and able to comply with all study procedures and restrictions
* Participant understands the study procedures and agrees to participate by providing written informed consent.

Exclusion Criteria:

* Participant with history or presence of any clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, endocrine, immunologic, dermatologic, neurological, psychiatric disease or disorder or any uncontrolled medical illness which in the opinion of the investigator would jeopardize the safety of the participant, interfere with study assessments, or impact the validity of the study results
* Participant with a history or family history of additional risk factors for Torsade de Pointe (TdP)
* Participant with a marked prolongation of ECG intervals, including QTcF >450 milliseconds (msec), PR >200 msec, or QRS >120 msec
* Participant with resting heart rate of <45beats per minute (bpm) or >100 bpm
* Participant with clinically significant abnormal ECG results
* Participant who uses medications that could prolong the QT/QTc interval
* Participant taking medications/dietary supplements that are highly dependent on cytochrome (CYP)3A for clearance and cannot undergo dose modification upon co-administration with strong CYP3A inhibitors
* Participant using any strong CYP3A inhibitor/inducer or any other medications prohibited per protocol
* Participant who is receiving testosterone within 40 days prior to study start
* Participant with a positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, or hepatitis C antibody
* Participant with a positive test result for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) viral RNA test, either asymptomatic or present with symptoms of Coronavirus disease 2019 (COVID-19)
* Participant who has travelled abroad within 3 months prior to the screening visit or plans to travel abroad during the study
* Participant who has had a major surgery within the last 28 days prior to Screening
* Participant who received any investigational product within 30 days prior to Screening
* Participant who has a known or suspected allergy, or sensitivity to study products, or any of its ingredient(s), or to moxifloxacin
* Intolerance to repeated venipuncture or inability to swallow capsules
* Donation of blood within 56 days or plasma within 14 days prior to Screening or plans to donate during the entire study period
* Positive alcohol test and/or positive drugs of abuse screen or reports of a history of substance or alcohol abuse within 1 year prior to Screening
* Female participant who is pregnant, breastfeeding, or is planning to become pregnant during the entire study period
* Male participant with pregnant partner.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected Change from Baseline in Cardiac QT Interval Corrected by Fridericia's Formula (QTcF) | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period

SECONDARY OUTCOMES:
Change from Baseline in Cardiac QTcF | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Change from Baseline in Heart Rate (HR) | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Placebo-corrected Change from Baseline in HR | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Change from Baseline in Cardiac PR Interval | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Placebo-corrected Change from Baseline in Cardiac PR Interval | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Change from Baseline in Cardiac QRS Intervals | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Placebo-corrected Change from Baseline in Cardiac QRS Intervals | Before dosing (Baseline) through 24 hours after the final dose on Day 5 in each treatment period
Number of Participants with a Categorical Outlier in QTcF | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Number of Participants with a Categorical Outlier in HR | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Number of Participants with a Categorical Outlier in PR Interval | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Number of Participants with a Categorical Outlier in QRS Intervals | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Number of Participants with a Treatment-emergent Change of T-wave Morphology | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Number of Participants with a Treatment-emergent Presence of U-waves | Up to Day 6 in each treatment period (through 24 hours after the final dose on Day 5 in each treatment period)
Maximum Plasma Concentration (Cmax) of Relacorilant, Metabolites of Relacorilant, and Moxifloxacin | Before dosing and at 0.5, 1, 1,5, 2, 3, 4, 6, 8, 12, 16, and 24 hours after dosing on Day 1 and 5 in each treatment period
Time to Reach Cmax (Tmax) of Plasma Relacorilant, Metabolites of Relacorilant, and Moxifloxacin | Before dosing and at 0.5, 1, 1,5, 2, 3, 4, 6, 8, 12, 16, and 24 hours after dosing on Day 1 and 5 in each treatment period
Minimum Plasma Concentration (Cmin) of Relacorilant, Metabolites of Relacorilant, and Moxifloxacin | Before dosing on Day 5 of each treatment period
Area Under the Plasma-concentration Curve from Time Zero to Time of Last Measurable Concentration (AUClast) of Relacorilant, Metabolites of Relacorilant, and Moxifloxacin | Before dosing and at 0.5, 1, 1,5, 2, 3, 4, 6, 8, 12, 16, and 24 hours after dosing on Day 1 and 5 in each treatment period
Area Under the Plasma-concentration Curve from Time Zero to 24 Hours Postdose (AUC0-24) of Relacorilant, Metabolites of Relacorilant, and Moxifloxacin | Before dosing and at 0.5, 1, 1,5, 2, 3, 4, 6, 8, 12, 16, and 24 hours after dosing on Day 1 and 5 in each treatment period
Number of Participants with One or More Adverse Events | Up to Day 6 in each treatment period (up to 51 days)
Number of Participants Discontinued From Study Treatment due to an Adverse Event | Up to Day 6 of each treatment period (up to 51 days)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Single Site, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No